CLINICAL TRIAL: NCT06827834
Title: A Prospective Longitudinal Study of Spinal Cord Lesions in Multiple Sclerosis: MRI Monitoring and Prognostic Factors for Active Disease
Brief Title: Spinal Cord Monitoring in Multiple Sclerosis
Acronym: MSpine
Status: Recruiting | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: Z2023148
Record Dates: First submitted 2025-01-27; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: spinal cord; mri; biomarkers; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Multiple sclerosis (MS) is the most common demyelinating disease of the central nervous system and the most common cause of non-traumatic neurological disability in young adults. Magnetic resonance imaging (MRI) is the most important paraclinical investigation used in the diagnosis and monitoring of the disease. In the past years, spinal cord MRI has improved significantly and has become an important part of the diagnostic workup for MS. Presently, follow-up imaging of the spinal cord is only performed when spinal cord related symptoms occur. However, there is increasing evidence that asymptomatic spinal cord lesions can occur, independently of brain disease activity. Despite these cord lesions being asymptomatic, they impact disability accrual in the long term. Although this might be an imaging marker for monitoring and treatment, it is not yet applied in the clinical setting.

The investigators will prospectively collect spinal cord MRI data (in addition to routine brain MRI), and blood-based biomarkers (plus cerebral spinal fluid markers, if available), in recently diagnosed MS patients, to address the following research questions:

* What is the incidence of asymptomatic spinal cord lesions in patients commencing DMT?
* And in the absence of radiological progression on brain imaging, how frequently do asymptomatic spinal cord lesions occur? In other words, how often is disease activity solely proven by spinal cord MRI and what is the number-needed-to-scan?
* A secondary objective is to investigate which patients are predisposed to developing new spinal cord lesions during follow-up in the early stages of the disease. For this question, factors such as cerebrospinal fluid (CSF) profiles, B-cell composition in blood, soluble blood markers, and clinical features will be focused on.

DETAILED DESCRIPTION:
The investigators aim to prospectively collect spinal cord MRI data (in addition to routine brain MRI), in recently diagnosed MS patients, to address the following research questions:

What is the incidence of asymptomatic spinal cord lesions in patients commencing DMT?

And in the absence of radiological progression on brain imaging, how frequently do asymptomatic spinal cord lesions occur? In other words, how often is disease activity solely proven by spinal cord MRI and what is the number-needed-to-scan?

1. What is the incidence of asymptomatic spinal cord lesions in patients commencing DMT?
2. In the absence of radiological progression on brain imaging, how frequently do asymptomatic spinal cord lesions occur? In other words, how often is disease activity solely proven by spinal cord MRI and what is the number-needed-to-scan?

Hypothesis: The hypothesis is that the detected incidence of asymptomatic cord lesions independent of brain MRI activity will be higher than the approximately 10% per year reported in retrospective studies.

A secondary objective is to investigate which patients are predisposed to developing new spinal cord lesions during follow-up in the early stages of the disease. For this question, factors such as cerebrospinal fluid (CSF) profiles, B-cell composition in blood, soluble blood markers, and clinical features will be focused on.

2. What subgroups are prone to new spinal cord lesions at follow-up in early disease? In particular:

* Can disease activity on spinal cord MRI be predicted by baseline CSF profiles, i.e. is there an association between intrathecal IgM/IgG synthesis, number of oligoclonal bands and/or kappa free light chains at baseline and formation of new spinal cord lesions at follow-up?
* Is there an association between low number of transitional B cells in blood at baseline and formation of new spinal cord lesions?
* Is there an association between soluble blood markers and other blood biomarkers at baseline and formation of new spinal cord lesions at follow-up?
* What subtype of clinical presentation or certain physical complaints are associated with new spinal cord lesions during follow-up?

Hypothesis: The hypothesis is that more new spinal cord lesions occur in patients with CSF profile positive for intrathecal IgM, IgG synthesis and higher number oligoclonal bands, a low number of transitional B cells at baseline, a low number of CD56bright NK cells, high levels of activating sICPs and low levels of inhibitory sICPs at baseline, and/or a presenting syndrome of optic neuritis or myelitis.

To investigate the research questions, MS patients will be enrolled from five Dutch MS centres in an observational study with a follow-up of 27 months. Patients will be asked to participate when they are being screened for DMT initiation and given 7 days to consider. Informed consent will be obtained by a doctor, part of the research team. Next to routine regular follow-up with brain MRI and outpatient clinic visits, patients will receive spinal cord MRI and a structured registration of clinical parameters and collection of blood samples. Towards the end of follow-up, it will be evaluated whether starting an extension study is of additional value.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old
* Patients diagnosed with relapsing-remitting MS (≤5 years of first clinical event)
* Treatment-naïve patients starting (currently in the Netherlands approved) DMT

Exclusion Criteria:

* Patients who presented first clinical event more than five years ago
* Patients who have already started DMT
* Patients who are incapable of giving informed consent
* Patients who are unable to undergo local MRI scan, due to for instance
* Physical problems, for instance due to size/obesity (not fitting in regular MRI scanner), not being able to lie flat for extended periods of time (e.g. due to pain, shortness of breath)
* Due to claustrophobia
* Patients who have contraindications for MRI scan, for instance
* Due to MRI-unsafe or non-compatible implanted material/devices, such as pacemakers or ocular metal splinters
* Patients who are pregnant at inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of treatment-naïve relapsing-remitting MS patients, early in the disease course (within 5 years of first clinical event) between 18 - 65 years old, where a first DMT is initiated.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Spinal cord lesion count | 27 months

SECONDARY OUTCOMES:
Brain MRI acitivity | 27 months
  Number of new (new T2, T1 gadolinium-enhancing) and expanding lesions
Expanded disability status scale (EDSS) | 27 months
  Measured at 3, 15 and 27 months
Timed 25 foot walk test | 27 months
  Measured at 3, 15 and 27 months
Nine hole peg test | 27 months
  Measured at 3, 15 and 27 months
No evidence of disease activity | 27 months
  Composite outcome: no relapses, no progression independent of relapse activity, no new lesions on brain or spinal cord MRI
Biomarkers neuronal damage | 27 months
  Neurofilament light chain (Nfl) and glial fibrillary acidic protein (GFAP)
Lower urinary tract symptoms | 27 months
  * For females: International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Module (ICIQ-FLUTS)
  * For males: International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms Module (ICIQ-MLUTS)

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Rijnstate, Arnhem, Gelderland
  - Zuyderland Medisch Centrum, Geleen, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Albert Schweitzer ziekenhuis, Dordrecht, South Holland
  - Erasmus MC, Rotterdam, South Holland

REFERENCES:
- [Background] Di Sabatino E, Gaetani L, Sperandei S, Fiacca A, Guercini G, Parnetti L, Di Filippo M. The no evidence of disease activity (NEDA) concept in MS: impact of spinal cord MRI. J Neurol. 2022 Jun;269(6):3129-3135. doi: 10.1007/s00415-021-10901-2. Epub 2021 Nov 24. PMID 34820734
- [Background] Kreiter D, Spee R, Merry A, Hupperts R, Gerlach O. Effect of disease-modifying treatment on spinal cord lesion formation in multiple sclerosis: A retrospective observational study. Mult Scler Relat Disord. 2023 Nov;79:104994. doi: 10.1016/j.msard.2023.104994. Epub 2023 Sep 4. PMID 37683557
- [Background] Brownlee WJ, Altmann DR, Alves Da Mota P, Swanton JK, Miszkiel KA, Wheeler-Kingshott CG, Ciccarelli O, Miller DH. Association of asymptomatic spinal cord lesions and atrophy with disability 5 years after a clinically isolated syndrome. Mult Scler. 2017 Apr;23(5):665-674. doi: 10.1177/1352458516663034. Epub 2016 Aug 6. PMID 27481210
- [Background] Granella F, Tsantes E, Graziuso S, Bazzurri V, Crisi G, Curti E. Spinal cord lesions are frequently asymptomatic in relapsing-remitting multiple sclerosis: a retrospective MRI survey. J Neurol. 2019 Dec;266(12):3031-3037. doi: 10.1007/s00415-019-09526-3. Epub 2019 Sep 7. PMID 31494713
- [Background] Zecca C, Disanto G, Sormani MP, Riccitelli GC, Cianfoni A, Del Grande F, Pravata E, Gobbi C. Relevance of asymptomatic spinal MRI lesions in patients with multiple sclerosis. Mult Scler. 2016 May;22(6):782-91. doi: 10.1177/1352458515599246. Epub 2015 Oct 12. PMID 26459149